CLINICAL TRIAL: NCT05766462
Title: Utilization of Personalized Pacing to Improve Quality of Life in Sinus Node Dysfunction Patients
Brief Title: Allometric-Pace Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Allometric-Pace Study
Record Dates: First submitted 2023-02-20; First posted 2023-03-13 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-05

CONDITIONS: Sinus Node Dysfunction
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PLR group: The pacemaker lower rate of PLR group will be set as 75 bpm and might be adjusted according to physician diagnosis based on patients situation.
  Interventions: Other: Pacemaker lower rate setting
- control group: The pacemaker lower rate of control group will be set as 60 bpm.

INTERVENTIONS:
Other: Pacemaker lower rate setting — Pacemaker lower rate is set by physician and may be adjusted according to the physician diagnosis.
  Groups: PLR group

SUMMARY:
The goal of this observational study is to improve quality of life in sinus node dysfunction patients by utilizing allometric lower rate pacing (or called personalized lower rate, PLR) in standard commercially available dual-chamber pacemakers.

The primary objective is to achieve a significant improvement in patients' quality of life with use of PLR pacing in comparison with the control group with nominal lower rate in patients with implanted dual-chamber pacemaker.

The secondary objectives are to assess cardiac functional changes in echocardiography of ventricular mechanical performance with a PLR pacing in comparison with the control group with nominal lower rate, and to assess the viability of using elevated blood pressure as a marker for undetected bradycardia and providing allometric rate to correct bradycardia-related increase in arterial systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients are at age of equal to or more than 60 years old
* Patients have plan to implant dual-chamber pacemaker
* Resting sinus heart rate is equal or less than 60 bpm, or average heart rate detected through 24-hour dynamic electrocardiogram is equal or less than 60 bpm
* Patients have diagnosis of SND. If patients have both sinus node dysfunction and AV block, conduction system pacing shall be available
* Patients have a history of hypertension, two times of blood pressure measurements at office visit are equal to or more than 130 mmHg in systolic blood pressure, diastolic pressure is equal or less than 80 bpm

Exclusion Criteria:

* Patients have or possible concomitant a diagnosis of heart failure, either reduced EF or preserved EF
* Patients have persistent or chronic atrial fibrillation or clinically significant paroxysmal atrial fibrillation
* Previously diagnosed with a history of organic heart disease: including congenital heart disease, coronary heart disease, old myocardial infarction, dilated cardiomyopathy, hypertrophic cardiomyopathy, cardiac amyloidosis, long QT syndrome, etc.
* Patients have a known secondary cause of hypertension
* Patients have hospitalization of a hypertensive emergency in the previous year
* Patients have a history of renal disease or renal-artery diseases
* Severe hepatic or renal dysfunction
* Active acute infection
* Patients cannot submit a signed informed consent form
* Patients are pregnant or plan to be pregnant during study period
* Patients participate in another study that will confound this study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The three sites locate in the north, west and south of China respectively and are all Tertiary A hospitals. This study will enroll 70 subjects who meet all the inclusion and exclusion criteria from the in-patients from the three hospitals.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Life quality measurement | Within three months after the surgery
  SF-36 questionnaire score will be used as the criteria.

SECONDARY OUTCOMES:
Cardiac functional changes | Within three months after the surgery
  LVEF will be measured
To assess the correlation of elevated blood pressure and bradycardia. | Within three months after the surgery
  24 hour ambulatory blood pressure will be measured.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassil G, Zarzoso M, Noujaim SF. Allometric scaling of electrical excitation and propagation in the mammalian heart. J Theor Biol. 2017 Apr 21;419:238-242. doi: 10.1016/j.jtbi.2016.09.024. Epub 2016 Sep 26. PMID 27686596
- [Background] Infeld M, Avram R, Wahlberg K, Silverman DN, Habel N, Lustgarten DL, Pletcher MJ, Olgin JE, Marcus GM, Meyer M. An approach towards individualized lower rate settings for pacemakers. Heart Rhythm O2. 2020 Dec;1(5):390-393. doi: 10.1016/j.hroo.2020.09.004. Epub 2020 Oct 6. No abstract available. PMID 33604585
- [Background] Infeld M, Wahlberg K, Cicero J, Meagher S, Habel N, Muthu Krishnan A, Silverman DN, Lustgarten DL, Meyer M. Personalized pacing for diastolic dysfunction and heart failure with preserved ejection fraction: Design and rationale for the myPACE randomized controlled trial. Heart Rhythm O2. 2021 Dec 7;3(1):109-116. doi: 10.1016/j.hroo.2021.11.015. eCollection 2022 Feb. PMID 35243443